CLINICAL TRIAL: NCT00984282
Title: A Double-Blind Randomized Phase III Study Evaluating the Efficacy and Safety of Sorafenib Compared to Placebo in Locally Advanced/Metastatic RAI-Refractory Differentiated Thyroid Cancer
Brief Title: Nexavar® Versus Placebo in Locally Advanced/Metastatic RAI-Refractory Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14295; 2009-012007-25 (EudraCT Number)
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Thyroid Neoplasms
Keywords: RAI-Refractory; Differentiated; Follicular; Papillary; Hurthle
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Participants received 2 tablets of Sorafenib (2×200 mg) orally twice daily (12 hours apart without food), 28 days comprise a cycle
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Placebo (Placebo Comparator): Participants received 2 tablets of Sorafenib-matching placebo orally twice daily (12 hours apart without food), 28 days comprise a cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 400 mg will be administered orally, twice daily (approximately every 12 hours).
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Placebo — Placebo (2 tablets) will be administered orally, twice daily (approximately every 12 hours).
  Arms: Placebo

SUMMARY:
Trial of sorafenib versus placebo in the treatment of locally advanced or metastatic differentiated thyroid cancer refractory to radioiodine

DETAILED DESCRIPTION:
Eligible subjects were randomized 1:1 to sorafenib 800 mg daily or matching placebo. Progression was assessed every 8 weeks by modified RECIST criteria. Subjects had the option to unblind study treatment after progression and to receive open label sorafenib regardless of initial treatment assignment. Following discontinuation of study treatment, subjects were followed for survival every 3 months in long-term follow-up. Subjects who terminated study treatment (either double only or double blind and open label) for reasons other than death, lost to follow-up or consent withdrawn entered long-term follow up

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic differentiated thyroid cancer (papillary, follicular and Hurthle cell)
* Poorly differentiated and other thyroid variants (e.g. insular, tall cell, etc.) are eligible provided that the histology has no medullary differentiation nor anaplastic features
* Progression within 14 months (RECIST [Response Evaluation Criteria in Solid Tumors] should be used as a basis for the assessment of disease progression)
* RAI (radioactive iodine) refractory

Exclusion Criteria:

* Histologic subtypes of thyroid cancer other than differentiated (i.e. like anaplastic and medullary carcinoma, lymphoma or sarcoma)
* Prior anti-cancer treatment with tyrosine kinase inhibitors, monoclonal antibodies (licensed or investigational) that target VEGF (vascular endothelial growth factor) or VEGF Receptors or other targeted agents
* Prior anti-cancer treatment for thyroid cancer with use of chemotherapy (low dose chemotherapy for radiosensitization is allowed) or Thalidomide or any of its derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2009-10-15 (Actual); Primary Completion 2012-08-31 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (71):
- United States (13):
  - Los Angeles, California
  - Stanford, California
  - New Haven, Connecticut
  - Atlanta, Georgia
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Seattle, Washington
- Vienna, Austria
- Bruxelles - Brussel, Belgium
- Sofia, Bulgaria
- China (6):
  - Guangzhou, Guangdong
  - Beijing
  - Chengdu
  - Hangzhou
  - Shanghai
  - Tianjin
- Odense C, Denmark
- France (8):
  - Angers
  - Bordeaux
  - Caen
  - Lille
  - Lyon
  - Marseille
  - Paris
  - Villejuif
- Germany (6):
  - Erlangen, Bavaria
  - München, Bavaria
  - Würzburg, Bavaria
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Leipzig, Saxony
- Italy (7):
  - Napoli, Campania
  - Genoa, Liguria
  - Milan, Lombardy
  - Catania, Sicily
  - Pisa, Tuscany
  - Siena, Tuscany
  - Perugia, Umbria
- Japan (3):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Koto-ku, Tokyo
- Netherlands (2):
  - Groningen
  - Leiden
- Poland (3):
  - Gliwice
  - Poznan
  - Warsaw
- Obninsk, Russia
- Riyadh, Saudi Arabia
- South Korea (3):
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Daejeon
  - Seoul
- Spain (2):
  - Majadahonda, Madrid
  - Barcelona
- Sweden (4):
  - Gothenburg
  - Linköping
  - Lund
  - Stockholm
- United Kingdom (8):
  - Aberdeen, Aberdeenshire
  - Cardiff
  - Glasgow
  - Leeds
  - London
  - Manchester
  - Newcastle upon Tyne
  - Sutton

REFERENCES:
- [Result] Worden F, Fassnacht M, Shi Y, Hadjieva T, Bonichon F, Gao M, Fugazzola L, Ando Y, Hasegawa Y, Park DJ, Shong YK, Smit JW, Chung J, Kappeler C, Meinhardt G, Schlumberger M, Brose MS. Safety and tolerability of sorafenib in patients with radioiodine-refractory thyroid cancer. Endocr Relat Cancer. 2015 Dec;22(6):877-87. doi: 10.1530/ERC-15-0252. PMID 26370187
- [Result] Brose MS, Nutting CM, Jarzab B, Elisei R, Siena S, Bastholt L, de la Fouchardiere C, Pacini F, Paschke R, Shong YK, Sherman SI, Smit JW, Chung J, Kappeler C, Pena C, Molnar I, Schlumberger MJ; DECISION investigators. Sorafenib in radioactive iodine-refractory, locally advanced or metastatic differentiated thyroid cancer: a randomised, double-blind, phase 3 trial. Lancet. 2014 Jul 26;384(9940):319-28. doi: 10.1016/S0140-6736(14)60421-9. Epub 2014 Apr 24. PMID 24768112
- [Result] Brose MS, Nutting CM, Sherman SI, Shong YK, Smit JW, Reike G, Chung J, Kalmus J, Kappeler C, Schlumberger M. Rationale and design of decision: a double-blind, randomized, placebo-controlled phase III trial evaluating the efficacy and safety of sorafenib in patients with locally advanced or metastatic radioactive iodine (RAI)-refractory, differentiated thyroid cancer. BMC Cancer. 2011 Aug 11;11:349. doi: 10.1186/1471-2407-11-349. PMID 21834960
- [Derived] Brose MS, Schlumbeger M, Jeffers M, Kappeler C, Meinhardt G, Pena CEA. Analysis of Biomarkers and Association With Clinical Outcomes in Patients With Differentiated Thyroid Cancer: Subanalysis of the Sorafenib Phase III DECISION Trial. Clin Cancer Res. 2019 Dec 15;25(24):7370-7380. doi: 10.1158/1078-0432.CCR-18-3439. Epub 2019 Sep 26. PMID 31558473
- [Derived] Capdevila J, Matos I, Mancuso FM, Iglesias C, Nuciforo P, Zafon C, Palmer HG, Ogbah Z, Muinos L, Hernando J, Villacampa G, Pena CE, Tabernero J, Brose MS, Schlumberger M, Vivancos A. Identification of Expression Profiles Defining Distinct Prognostic Subsets of Radioactive-Iodine Refractory Differentiated Thyroid Cancer from the DECISION Trial. Mol Cancer Ther. 2020 Jan;19(1):312-317. doi: 10.1158/1535-7163.MCT-19-0211. Epub 2019 Sep 20. PMID 31540966
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 556 screened participants, 137 failed screening, 207 were randomized to receive sorafenib, 210 were randomized to placebo.
Groups:
- DB Sorafenib First, Then Option of OL Sorafenib Treatment: Double-blind period: Participants received 2 tablets of Sorafenib (2×200 mg) orally twice daily (12 hours apart without food), 28 days comprise a cycle. Open-label (OL) period: Participants received 2 tablets of Sorafenib (2×200 mg) orally twice daily (12 hours apart without food), 28 days comprise a cycle.
- DB Placebo First, Then Option of OL Sorafenib Treatment: Double-blind period: participants received matching placebo tablets orally twice daily, 28 days comprised a cycle. Open-label (OL) period: participants on placebo who switched to sorafenib, received sorafenib 400 mg (2 x 200 mg) orally twice daily, 28 days comprise a cycle.
Period: Double Blind Treatment
Arm/Group | DB Sorafenib First, Then Option of OL Sorafenib Treatment | DB Placebo First, Then Option of OL Sorafenib Treatment
Started | 207 | 210
Received Treatment | 207 (Subjects at Risk/Safety Population - in RG1 (RG= Reporting Group for Safety Data)) | 209 (Subjects at Risk/Safety Population - in RG2 (RG= Reporting Group for Safety Data))
Completed | 103 | 172
Not Completed | 104 | 38
Not completed — Adverse Event | 40 | 6
Not completed — Progression, recurrence or relapse | 25 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Noncompliance with study medication | 3 | 0
Not completed — Progression by clinical judgment | 2 | 0
Not completed — Withdrawal by Subject | 13 | 18
Not completed — Lost to Follow-up | 3 | 0
Not completed — Death | 8 | 4
Not completed — Not treated | 0 | 1
Not completed — Switched to commercial drug | 6 | 1
Not completed — protocol driven decision point | 1 | 1
Not completed — Radiological and clinical progression | 0 | 1
Not completed — Transferred to treat. continuation study | 2 | 1
Period: Open-label Treatment
Arm/Group | DB Sorafenib First, Then Option of OL Sorafenib Treatment | DB Placebo First, Then Option of OL Sorafenib Treatment
Started | 86 | 161
Received Treatment | 86 (Subjects at Risk/Safety Population - in RG3 (RG= Reporting Group for Safety Data)) | 161 (Subjects at Risk/Safety Population - in RG4 (RG= Reporting Group for Safety Data))
Completed | 0 | 0
Not Completed | 86 | 161
Not completed — Adverse Event | 20 | 30
Not completed — Withdrawal by Subject | 6 | 21
Not completed — Death | 7 | 15
Not completed — Progression, recurrence or relapse | 40 | 82
Not completed — Lost to Follow-up | 1 | 1
Not completed — Patient convenience | 1 | 0
Not completed — Non-compliant with study medication | 1 | 0
Not completed — Target lesion removed | 0 | 1
Not completed — Protocol driven decision point | 1 | 1
Not completed — Transferred to treat. continuation study | 2 | 3
Not completed — Switched to commercial drug | 6 | 7
Not completed — Physician Decision | 1 | 0
Period: Long Term Follow-up
Arm/Group | DB Sorafenib First, Then Option of OL Sorafenib Treatment | DB Placebo First, Then Option of OL Sorafenib Treatment
Started | 72 (Participants entered long-term follow-up if terminated double-blind or open-label periods) | 124 (Participants entered long-term follow-up if terminated double-blind or open-label periods)
Completed | 3 | 4
Not Completed | 69 | 120
Not completed — Withdrawal by Subject | 8 | 14
Not completed — Death | 27 | 68
Not completed — Lost to Follow-up | 3 | 6
Not completed — Protocol driven decision point | 25 | 26
Not completed — Transferred to treat. continuation study | 2 | 3
Not completed — Switched to commercial drug | 4 | 2
Not completed — Disease prog., recurrence or relapse | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Total
Number analyzed (Participants) | 207 | 210 | 417
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (11.2) | 62.0 (11.7) | 61.8 (11.4)
Age, Customized [Count of Participants; unit: Participants]
  < 60 years | 80 | 81 | 161
  >= 60 years | 127 | 129 | 256
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 115 | 218
  Male | 104 | 95 | 199
Geographic region [Count of Participants; unit: Participants]
  Europe | 124 | 125 | 249
  North America | 36 | 36 | 72
  Asia | 47 | 49 | 96
ECOG (Eastern Cooperative Oncology Group) performance status [Count of Participants; unit: Participants] — The ECOG PS required for the study was 0 (fully active), 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), or 2 (ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  Participants
    Missing | 1 | 1 | 2
    0 | 130 | 129 | 259
    1 | 69 | 74 | 143
    2 | 7 | 6 | 13
Site of target/nontarget lesions at baseline - organ class [Number; unit: Participants] — Participants could have had more than one site.
  Participants
    Lung | 178 | 181 | 359
    Lymph node | 113 | 101 | 214
    Bone | 57 | 56 | 113

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Central Assessment Incl. Clinical Progression Due to Bone Irradiation
Description: PFS=time from randomization to first observed disease progression (radiological according to central assessment or clinical due to bone irradiation, whichever is earlier), or death due to any cause, if death occurred before progression. Progression was assessed by RECIST criteria, version 1.0, modified for bone lesions. PFS for participants without disease progression or death at the time of analysis or unblinding were censored at the last date of tumor assessment before unblinding. Participants with no tumor evaluation after baseline were censored at Day 1. PD (Progression Disease)=At least a 20% increase in sum of longest diameters (LD) of measured lesions taking as reference the smallest sum LD on study since the treatment started or the appearance of 1 or more new lesions. New lesions also constituted PD. In exceptional circumstances, unequivocal progression of a nonmeasured lesion may have been accepted as evidence of disease progression in participants with measurable disease.
Time Frame: Final analysis to be performed when approximately 267 progression-free survival events (centrally assessed) had occurred, study duration approximately three years
Population: Full Analysis Set (FAS). The primary population for efficacy analysis was the FAS. The FAS was identical to the intent-to-treat (ITT) population, which was defined as all randomized participants. Participants were analyzed as randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 207 | 210
Days | 329 [278 to 393] | 175 [160 to 238]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; The two treatment groups were compared using a stratified one-sided log rank test with an overall alpha of 0.01 stratified by age group and region. The null hypothesis that both treatment arms have the same PFS distribution will be tested against the alternative hypothesis that the distribution of PFS times in the sorafenib arm is different from the control arm according to the Lehmann alternative, which is equivalent to the assumption of proportional hazards of the treatment arms; Test type: Superiority or Other; p < 0.0001, Log Rank — stratified by age group (< 60 years, >= 60 years) and region (Europe, North-America, Asia)
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; Regression, Cox; stratified by age group and region; Hazard Ratio (HR) = 0.587, 95% CI 2-sided [0.454 to 0.758]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time (days) from date of randomization to date of death due to any cause. Subjects still alive at the time of analysis were censored at their date of last contact. Since the median value could not be estimated due to censored data, the percentage of participants who died is presented.
Time Frame: From randomization of the first subject until the database cut-off (30 AUG 2017), study duration approximately eight years
Population: Full Analysis Set (FAS)
Measure: Number; unit: Percentage of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 207 | 210
Percentage of participants | 52.7 | 54.8
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.2892, Log Rank; stratified by age group and region
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; Regression, Cox; stratified by age group and region; Hazard Ratio (HR) = 0.928, 95% CI 2-sided [0.713 to 1.208]

3. Secondary Outcome: Time to Progression (TTP) Based on Central Assessment Incl. Clinical Progression Due to Bone Irradiation
Description: Time to progression was defined at the time (days) from randomization to progression (based on central assessment [radiological and clinical progression due to bone irradiation])
Time Frame: From randomization of the first subject until the database cut-off (31 Aug 2012), study duration approximately three years
Population: FAS
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 207 | 210
Days | 337 [283 to 451] | 175 [160 to 238]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank; stratified by age group and region
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; Regression, Cox; stratified by age group and region; Hazard Ratio (HR) = 0.557, 95% CI 2-sided [0.429 to 0.724]

4. Secondary Outcome: Disease Control Rate (DCR) Based on Central Assessment
Description: Disease control rate was defined as the proportion of subjects whose best response was complete response (CR), partial response (PR), or stable disease (SD). Per Response Evaluation Criteria in Solid Tumors (RECIST) criteria, CR and PR were to be confirmed by another scan at least 4 weeks later; SD had to be documented at least 4 weeks after date of randomization. CR = Disappearance of all clinical and radiological evidence of tumor (both target and no-target). PR = At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum. SD = steady state of disease which is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: as for outcome 3
Population: Per protocol set (PPS). A participant was included in the PPS if he/she was randomized and was evaluable for tumor response based on imaging data, had exposure to study medication, and had no major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 196 | 201
Percentage of participants | 86.2 [80.6 to 90.7] | 74.6 [68.0 to 80.5]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.0015, Cochran-Mantel-Haenszel — stratified by age group and region; Difference of response rates = 11.7, 95% CI 2-sided [3.9 to 19.4] — Difference of disease control rates sorafenib minus placebo. Cochran-Mantel-Haenszel confidence interval stratified by age group and region

5. Secondary Outcome: Response Rate Based on Central Assessment
Description: Response rate was defined as the proportion of subjects whose best response was CR or PR. Per RECIST, CR and PR was to be confirmed by another scan at least 4 weeks later. CR = Disappearance of all clinical and radiological evidence of tumor (both target and no-target). PR = At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum.
Time Frame: as for outcome 3
Population: PPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 196 | 201
Percentage of participants | 12.24 [8.01 to 17.67] | 0.5 [0.01 to 2.74]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — stratified by age group and region; Difference in response rate = 11.8, 95% CI 2-sided [7.0 to 16.5] — Difference of response rates sorafenib minus placebo. Cochran-Mantel-Haenszel confidence interval stratified by age group and region

6. Secondary Outcome: Duration of Response (DOR) Based on Central Assessment
Description: Duration of response was defined as the time from the first documented objective response of PR or CR, whichever was noted earlier, to disease progression or death (if death occurred before progression was documented). CR = Disappearance of all clinical and radiological evidence of tumor (both target and no-target). PR = At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum.
Time Frame: as for outcome 3
Population: FAS - responders only
Measure: Median (Full Range); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 24 | 1
Days | 309 [226 to 505] | NA [NA to NA] — only one subject with PR

7. Secondary Outcome: Maximum Percent Reduction in Target Lesion Size Based on Central Assessment
Description: The magnitude of change from baseline in target lesion size in evaluable participants with scans was determined.
Time Frame: as for outcome 3
Population: PPS
Measure: Number; unit: Percentage of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 196 | 201
Percentage of participants
  Reduction ≥ 30% | 17.3 | 1.0
  Reduction ≥ 20% but < 30% | 15.3 | 1.5
  Reduction ≥ 10% but < 20% | 22.4 | 3.5
  Reduction > 0% but < 10% | 22.4 | 21.9
  Growth ≥ 0% | 12.8 | 62.7
  Not assessed | 9.7 | 9.5

8. Secondary Outcome: AUC(0-12h),ss (Area Under the Concentration Time Curve From Time 0 to 12 Hours at Steady State)
Description: Sorafenib AUC(0-12h),ss (area under the concentration time curve from time 0 to 12 hours at steady state) was estimated from the steady state plasma concentration.
Time Frame: A single pharmacokinetic plasma sample was collected at steady state (after 14 days of uninterrupted, unmodified sorafenib dosing)
Population: Pharmacokinetic (PK) analysis set=participants with PK data collected after 14 days of uninterrupted and unmodified dosing of sorafenib. If an interruption occurred within 14 days prior to the sample, no doses may be missed for 3 days prior to the sample, and no more than 3 doses could be missed 4 to 14 days prior to the sample collection date.
Measure: Geometric Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 113
mg*h/L | 75.4 (1.5)

ADVERSE EVENTS:
Time Frame: After signing the informed consent until the database cut-off 30 AUG 2017, study duration approximately eight years.
Description: Abbreviations used: Gastrointestinal (GI), Common Terminology Criteria for Adverse Events (CTCAE), Not Otherwise Specified (NOS), Absolute Neutrophil Count (ANC), Central Nervous System (CNS), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Cranial Nerve (CN), Range of Motion (ROM), Cerebrospinal Fluid (CSF), Genitourinary (GU).
Groups:
- Sorafenib (Double Blind Only): Reporting Group 1: Participants received 2 tablets of Sorafenib (2x200 mg) orally twice daily (12 hours apart without food), 28 days comprise a cycle. Data were collected from randomization to the end of double blind period
- Placebo (Double Blind Only): Reporting Group 2: Participants received 2 tablets of Sorafenib-matching placebo orally twice daily (12 hours apart without food), 28 days comprise a cycle. Data were collected from randomization to the end of double-blind period.
- Sorafenib, Open Label Only (Sorafenib Continued): Reporting Group 3: Participants on sorafenib who continued OL sorafenib treat., received sorafenib 400 mg (2 x 200 mg) orally twice daily, 28 days comprise a cycle. Data were collected from the start of OL period to the data cutoff on 31 Aug
- Placebo, Open Label Only (Switch to Sorafenib): Reporting Group 3: Participants on placebo who switched to sorafenib, received sorafenib 400 mg (2 x 200 mg) orally twice daily, 28 days comprise a cycle. Data were collected from the start of open label period to the data cutoff on 31 Aug 20
Arm/Group | Sorafenib (Double Blind Only) | Placebo (Double Blind Only) | Sorafenib, Open Label Only (Sorafenib Continued) | Placebo, Open Label Only (Switch to Sorafenib)
All-Cause Mortality (participants affected / at risk) | 71/207 | 25/209 | 38/86 | 90/161
Serious Adverse Events (participants affected / at risk) | 87/207 | 58/209 | 51/86 | 96/161
Other Adverse Events (participants affected / at risk) | 202/207 | 173/209 | 74/86 | 159/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (Double Blind Only) (N=207) | Placebo (Double Blind Only) (N=209) | Sorafenib, Open Label Only (Sorafenib Continued) (N=86) | Placebo, Open Label Only (Switch to Sorafenib) (N=161)
Blood - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (5)
Lymphatics - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrhythmia - Other (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cardiac general - Other (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (4)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular arrhythmia, Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Supraventricular arrhythmia, Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular arrhythmia, Supraventricular tachycardia (Cardiac disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Valvular heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia, Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocrine - Other (Endocrine disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular - Other (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic disc edema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 1 (1)
Fistula, GI, Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fistula, GI, Esophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GI - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (9) | 1 (1) | 1 (7) | 0 (0)
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis (functional/symptomatic), Trachea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction, GI, Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstruction, GI, Gallbladder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perforation, GI, Colon (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stricture, GI, Esophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcer, GI, Rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constitutional symptoms - Other (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Death not associated with CTCAE term, Death NOS (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Death not associated with CTCAE term, Disease progression NOS (General disorders) | 2 (2) | 2 (2) | 3 (3) | 9 (9)
Death not associated with CTCAE term, Multi-Organ Failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Death not associated with CTCAE term, Sudden death (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Flu-like syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
No code in CTCAE (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Not coded yet (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain, Abdomen NOS (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pain, Back (General disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Pain, Bone (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pain, Chest wall (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain, Chest/Thorax NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain, Dental/Teeth/peridontal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain, Extremity - limb (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain, Head/Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain, Joint (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain, Liver (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain, Lymph node (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain, Neuralgia/Peripheral nerve (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain, Pelvis (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain, Stomach (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain, Throat/Pharynx/Larynx (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain, Tumor pain (General disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Syndromes - Other (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor flare (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary - Other (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Liver dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Allergy - Other (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis, infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Documented clinically), Lung (Pneumonia) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Documented clinically), Soft tissue NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Documented clinically), Upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Documented clinically), Wound (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Infection with normal ANC, Anal/perianal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC, Bladder (urinary) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC, Blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC, Bone (Osteomyelitis) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC, Colon (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC, Kidney (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC, Lung (Pneumonia) (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Infection with normal ANC, Mediastinum NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC, Scrotum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC, Soft tissue NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC, Upper airway NOS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC, Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC, Wound (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC, Abdomen NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with unknown ANC, Appendix (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC, Bladder (urinary) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC, Blood (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC, Bronchus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC, Lung (Pneumonia) (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Infection with unknown ANC, Pleura (Empyema) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC, Prostate (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraop injury, Artery-aorta (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Intraop injury, Bone (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraop injury, Meninges (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraop injury, Neck NOS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraop injury, Thyroid (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intraop injury, Trachea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Extremity - upper (Function) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 2 (2) | 4 (4)
Lumbar spine ROM (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness, Extremity - lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, Extremity - upper (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 5 (6) | 4 (4)
Secondary malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (13) | 6 (6) | 4 (4) | 3 (3)
CNS ischemia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
CSF leak (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal nerve (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood Alteration, Anxiety (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood alteration, Depression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Neuropathy: Cranial, CN II Vision (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Fainting) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal - Other (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sexual - Other (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Airway obstruction, Larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Airway obstruction, Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Airway obstruction, Trachea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (8) | 2 (2) | 8 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (4) | 9 (13) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 3 (3)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CNS hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage - Other (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage pulmonary, Bronchopulmonary NOS (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage pulmonary, Bronchus (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage pulmonary, Larynx (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage pulmonary, Lung (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hemorrhage pulmonary, Respiratory tract NOS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI, Anus (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI, Colon (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hemorrhage, GI, Varices (rectal) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU, Urinary NOS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GU, Uterus (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis/Embolism (vascular access) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 (1) | 4 (4) | 2 (4) | 1 (1)
Vascular - Other (Vascular disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (Double Blind Only) (N=207) | Placebo (Double Blind Only) (N=209) | Sorafenib, Open Label Only (Sorafenib Continued) (N=86) | Placebo, Open Label Only (Switch to Sorafenib) (N=161)
Blood - Other (Blood and lymphatic system disorders) | 6 (6) | 6 (10) | 6 (20) | 10 (23)
Edema: Limb (Blood and lymphatic system disorders) | 13 (17) | 6 (7) | 8 (9) | 8 (11)
Hemoglobin (Blood and lymphatic system disorders) | 18 (24) | 10 (11) | 8 (9) | 26 (32)
Leukocytes (Blood and lymphatic system disorders) | 9 (13) | 4 (8) | 5 (6) | 8 (15)
Lymphopenia (Blood and lymphatic system disorders) | 7 (7) | 6 (8) | 1 (1) | 10 (13)
Platelets (Blood and lymphatic system disorders) | 8 (12) | 2 (2) | 3 (4) | 11 (15)
Hypertension (Cardiac disorders) | 85 (103) | 28 (35) | 10 (13) | 51 (57)
Anorexia (Gastrointestinal disorders) | 67 (89) | 12 (12) | 7 (9) | 48 (52)
Constipation (Gastrointestinal disorders) | 32 (38) | 18 (19) | 4 (4) | 27 (29)
Diarrhea (Gastrointestinal disorders) | 142 (226) | 32 (40) | 22 (26) | 96 (165)
Dry mouth (Gastrointestinal disorders) | 16 (16) | 8 (8) | 2 (2) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 14 (17) | 9 (9) | 5 (7) | 12 (14)
GI - Other (Gastrointestinal disorders) | 9 (11) | 4 (4) | 2 (3) | 10 (11)
Heartburn (Gastrointestinal disorders) | 10 (11) | 10 (10) | 1 (1) | 13 (14)
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 49 (58) | 7 (7) | 6 (14) | 41 (49)
Nausea (Gastrointestinal disorders) | 43 (55) | 25 (29) | 10 (12) | 52 (56)
Taste Alteration (Gastrointestinal disorders) | 16 (16) | 0 (0) | 1 (1) | 11 (12)
Vomiting (Gastrointestinal disorders) | 23 (36) | 13 (14) | 3 (3) | 18 (25)
Fatigue (General disorders) | 102 (132) | 52 (58) | 19 (23) | 68 (87)
Fever (General disorders) | 22 (30) | 10 (11) | 8 (10) | 21 (26)
Flu-like syndrome (General disorders) | 18 (32) | 10 (14) | 4 (5) | 11 (14)
Insomnia (General disorders) | 14 (16) | 6 (6) | 5 (5) | 16 (17)
Pain, Abdomen NOS (General disorders) | 30 (42) | 10 (10) | 6 (7) | 30 (38)
Pain, Back (General disorders) | 24 (28) | 21 (24) | 10 (11) | 15 (19)
Pain, Bone (General disorders) | 14 (21) | 18 (22) | 7 (12) | 12 (13)
Pain, Chest wall (General disorders) | 6 (8) | 3 (3) | 2 (2) | 9 (9)
Pain, Chest/Thorax NOS (General disorders) | 16 (20) | 5 (5) | 1 (1) | 17 (18)
Pain, Dental/Teeth/peridontal (General disorders) | 11 (15) | 4 (4) | 2 (2) | 11 (16)
Pain, Extremity - limb (General disorders) | 31 (49) | 19 (27) | 3 (3) | 28 (43)
Pain, Head/Headache (General disorders) | 38 (48) | 16 (17) | 3 (3) | 24 (29)
Pain, Joint (General disorders) | 20 (23) | 14 (19) | 5 (7) | 19 (25)
Pain, Muscle (General disorders) | 19 (23) | 15 (17) | 6 (6) | 11 (17)
Pain, Neck (General disorders) | 9 (10) | 6 (6) | 1 (1) | 9 (9)
Pain, Oral cavity (General disorders) | 7 (7) | 2 (2) | 0 (0) | 9 (11)
Pain, Other (General disorders) | 24 (30) | 16 (17) | 8 (13) | 27 (31)
Pain, Throat/Pharynx/Larynx (General disorders) | 21 (26) | 9 (11) | 1 (3) | 19 (24)
Weight loss (General disorders) | 102 (114) | 29 (30) | 29 (33) | 75 (85)
Rhinitis (Immune system disorders) | 9 (11) | 7 (10) | 2 (2) | 9 (10)
Infection - Other (Infections and infestations) | 22 (29) | 12 (19) | 8 (11) | 12 (17)
ALT (Metabolism and nutrition disorders) | 26 (29) | 9 (10) | 0 (0) | 15 (19)
AST (Metabolism and nutrition disorders) | 23 (26) | 5 (6) | 1 (2) | 11 (14)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 4 (4) | 5 (7) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 38 (54) | 11 (13) | 12 (21) | 30 (47)
Hypokalemia (Metabolism and nutrition disorders) | 14 (21) | 5 (6) | 4 (6) | 14 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (11) | 1 (1) | 0 (0) | 11 (12)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 79 (123) | 37 (50) | 21 (34) | 56 (101)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 19 (21) | 9 (9) | 7 (10) | 11 (16)
Dizziness (Nervous system disorders) | 14 (17) | 7 (8) | 1 (1) | 12 (13)
Mood Alteration, Anxiety (Nervous system disorders) | 7 (8) | 6 (6) | 0 (0) | 9 (10)
Neuropathy: sensory (Nervous system disorders) | 32 (42) | 13 (16) | 5 (6) | 21 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 (43) | 34 (39) | 9 (10) | 23 (28)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 31 (36) | 27 (32) | 10 (14) | 25 (32)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7) | 7 (11) | 7 (9)
Voice changes (Respiratory, thoracic and mediastinal disorders) | 25 (33) | 6 (6) | 2 (2) | 12 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 141 (155) | 18 (18) | 4 (4) | 96 (103)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 30 (56) | 6 (8) | 12 (14) | 31 (43)
Dry skin (Skin and subcutaneous tissue disorders) | 30 (36) | 12 (14) | 6 (7) | 17 (17)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 158 (223) | 20 (24) | 13 (15) | 109 (136)
Pruritus (Skin and subcutaneous tissue disorders) | 44 (52) | 22 (24) | 3 (6) | 21 (25)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 107 (166) | 25 (29) | 9 (10) | 67 (94)
Hemorrhage pulmonary, Nose (Vascular disorders) | 15 (17) | 2 (3) | 2 (2) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must discuss any publication with the sponsor prior to release and obtain written consent of the sponsor on the intended publication. He/she must send a draft manuscript of the publication 30 days in advance of submission in order to obtain approval prior to submission of the final version for publication. In case of a difference of opinion, the contents will be discussed in order to find a solution which satisfies both parties.